CLINICAL TRIAL: NCT02213016
Title: Evaluation of the Efficacy of Repetitive Transcranial Magnetic Stimulation on Cognitive, Anxiety and Depressive Symptoms in Patients Diagnosed With Major Depressive Disorder
Brief Title: Effectiveness of Repetitive Transcranial Magnetic Stimulation in Depressed Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Gabriela Armas Castañeda, Technical academic, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 141-2011
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Major Depression
Keywords: Stimulation magnetic transcranial, major depression, cognitive impairment
MeSH Terms: conditions — Depressive Disorder, Major; Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Transcranial magnetic stimulation (Sham Comparator): Sham repetitive Transcranial magnetic stimulation, 5 Hz, 5 sessions per week for three weeks: Total of 15 sessions.
  Interventions: Device: Sham Transcranial Magnetic Stimulation
- Transcraneal magnetic stimulation (Active Comparator): Active repetitive Transcranial magnetic stimulation, 5 Hz, 5 sessions per week for three weeks: Total of 15 sessions.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham Comparator (Sham Comparator): Sham repetitive Transcranial magnetic stimulation, 5 Hz, 2 sessions per week for 7 1/2 weeks: Total of 15 sessions.
  Interventions: Device: Sham Transcranial Magnetic Stimulation
- Active Comparator (Active Comparator): Active repetitive Transcranial magnetic stimulation, 5 Hz, 2 sessions per week for 7 1/2 weeks: Total of 15 sessions.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation
  Other Names: TMS device MagVenture model MagPro 100
  Arms: Active Comparator; Transcraneal magnetic stimulation
Device: Sham Transcranial Magnetic Stimulation
  Other Names: TMS device Magventure, model MagPro 100. COIL COOL-B65.
  Arms: Sham Comparator; Transcranial magnetic stimulation

SUMMARY:
The purpose of this study is to evaluate clinical efficacy (affective and cognitive) in patients with moderate depression between TMS over the left Dorsolateral Prefrontal Cortex (DLPFC) with simulated TMS, as well as clinical response when 5 sessions / week are applied vs. 2 sessions / week. All patients will receive 15 TMS sessions as initial treatment (active or sham) and respondents will participate in an TMS follow-up on the left DLPFC for three months.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled, parallel group clinical trial to evaluate the efficacy of two Transcranial Magnetic Stimulation (TMS) protocols in patients with major depressive disorder (MDD). 70 ambulatory patients with a MDD diagnosis from the Clinic at the Department of Psychiatry and Mental Health at the Universidad Nacional Autónoma de México (UNAM) will be included. All Patients will complete a total of 15 sessions of treatment in any of four groups: A group of patients will be randomly assigned to receive either 5 active TMS sessions or 2 sessions per week. Sham controls will also be randomly assigned to receive either 5 TMS sessions or 2 sessions per week. Afterwards, all participants will receive 2 sessions per month for a 3 month period. Depressive and anxiety symptoms will be evaluated at baseline, and every 5 TMS sessions during the acute treatment phase, and once at the end of a 3-month follow up. In addition, neuropsychological evaluations will be applied at baseline and at the end of the 15 session's treatment. Sessions will be applied with a MAG pro x 100 transcranial magnetic stimulator. Motor threshold will be set. Sessions will be applied over the left DLPFC at 5 Hz, 30 trains, 100%. Categorical variables will be described by percentages and frequencies. Continuous variables will be described by means and standard deviations. Treatment groups will be compared using Student's T test. Cognitive, anxiety and depressive symptom scale scores between treatment groups will be compared using repeated measures ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of major depressive disorder
* Having a greater or equal score to 18 points in the Ham-D scale at the moment of the initial evaluation
* Treatment free patients

Exclusion Criteria:

* Epilepsy or seizure risk record
* Carry metallic objects in the head (such as arterial clips, plates, screws), eye or brain

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Total scores on the Hamilton depression scale depression | After 15 sessions of treatment and at 3 months follow up

SECONDARY OUTCOMES:
Performance on the Wisconsin card sorting test | After 15 sessions of treatment and at 3 months follow-up

OTHER OUTCOMES:
Performance on stop signal task | After 15 sessions of treatment and at 3 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Mental Health, Faculty of Medicine, UNAM, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Unable to connect to PubMed to validate , last attempt on May 29, 2014 at 3:25 PM EDT
- [Derived] Armas-Castaneda G, Ricardo-Garcell J, Reyes JV, Heinze G, Salin RJ, Gonzalez JJ. Two rTMS sessions per week: a practical approach for treating major depressive disorder. Neuroreport. 2021 Dec 8;32(17):1364-1369. doi: 10.1097/WNR.0000000000001737. Epub 2021 Oct 28. PMID 34718252